CLINICAL TRIAL: NCT06752213
Title: Comparison of Manual Therapy and Auricular Vagus Nerve Stimulation in Chronic Low Back Pain: A Crossover Study
Brief Title: Comparison of Manual Therapy and Auricular Vagus Nerve Stimulation in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2797
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain; Pain
Keywords: pain; low back pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Vagus Nerve Stimulation; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve Stimulation (Experimental): Vagus nerve Stimulation
  Interventions: Device: Vagus nerve Stimulation; Other: Manual therapy
- Manual therapy (Experimental): manual therapy
  Interventions: Device: Vagus nerve Stimulation; Other: Manual therapy

INTERVENTIONS:
Device: Vagus nerve Stimulation — Vagus nerve Stimulation
Other: Manual therapy — Manual therapy

SUMMARY:
Especially in the elderly population, low back pain is a major health problem, causing great human costs, negatively affecting the quality of life and limiting the daily activities of individuals

ELIGIBILITY:
Inclusion criteria Patients aged 20-65 years with nonspecific chronic low back pain will be included in the study.

Exclusion criteria

* Cognitive impairment
* Severe osteoprosis
* Neurological deficit
* Being pregnant
* Operations on the lumbar region

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Muscle Endurance Assessment | 6 weeks
  Trunk Extensor Muscle Endurance To assess the endurance of the back extensor muscles, participants will lie prone on a table with their lower extremities stabilized. The trunk will hang off the table at the level of the anterior-superior iliac spine. At the start of the test, hands will be placed on a chair. Upon beginning, participants will position their arms alongside their trunk, holding their body parallel to the floor. The duration for which this position is maintained without breaking posture will be recorded in seconds.
  Trunk Flexor Muscle Endurance Participants will begin in a supine position with knees flexed and arms crossed over the chest. Starting from a 60-degree trunk flexion position, they will be asked to hold this posture. The legs will be stabilized at the knees, and the time the position is maintained will be recorded in seconds.
Autonomic Nervous System Assessment | 6 weeks
  Heart rate variability will be measured using the Polar H7 heart rate sensor with a chest strap and wrist monitor (Polar H7, Polar Electro Oy). The chest strap will be placed over the sternum, and heart rate data will be recorded before and after auricular VNS. This method is validated against electrocardiogram measurements.
Flamingo Balance Test | 6 weeks
  The Flamingo Balance Test, part of the Eurofit test battery, uses a stopwatch and a 50 cm-long, 4 cm-high, and 3 cm-wide wooden beam. Participants stand on their non-dominant leg on the beam, holding the opposite leg's knee in maximal flexion with the corresponding hand while focusing on a fixed point at eye level. The timer starts once the participant releases the examiner's hand and stops when balance is lost or the body touches the ground. The test is repeated three times, and the average score is recorded.
Modified Star Excursion Balance | 6 weeks
  Y-shape, with the anterior direction at 0° and the posteromedial and posterolateral directions set at 135° and 90° angles, respectively. Participants will stand on their dominant leg, maintaining balance while reaching with the non-dominant leg as far as possible in each direction. They will then return to the starting position. Four practice trials will be provided, followed by three test trials in each direction. The average of the test trials will be recorded.
Algometer | 6 weeks
  A digital algometer (Wagner Force Ten FDX 50 Wagner Instruments, Greenwich, CT) will be used to objectively assess pain threshold and tolerance. Measurements will be conducted on the most painful taut band within the trigger point identified during diagnostic evaluation. A 1 cm² disk probe will apply pressure until the participant signals the first sensation of pain by saying "stop."
Visual Analog Scale (VAS) | 6 weeks
  The VAS was used to assess pain intensity before and after treatment. Patients marked their pain level on a 10 cm line, with 0 representing no pain and 10 representing unbearable pain. The distance from the 0-point to the mark was measured in centimeters and recorded.
Oswestry Disability Index (ODI) | 6 weeks
  The Turkish version of the ODI is frequently used in clinical practice to evaluate functional disability in individuals with low back pain. The 10-item questionnaire assesses pain and daily living activities, with each item scored from 0 to 5. The total score is calculated using the formula: (Total score/Maximum score) × 100. Higher scores indicate greater disability.
Range of Motion and Mobility Assessment | 6 weeks
  Trunk flexion and extension ROM measurements will be performed using the Angles Video Goniometer app for iPhone™ (Angles app, © 2020 Nathaniel Joseph Cochran). For lumbar mobility evaluation, the modified Schober test and fingertip-to-floor distance (FTFD) test will be utilized.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazal GENÇ, Istanbul, None Selected, Turkey (Türkiye)